CLINICAL TRIAL: NCT02880813
Title: The Effects of Gastric or Duodenal Nutrient Infusion on Food Intake, Obesity and Comorbidities in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amy E Rothberg, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00106668
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric (Experimental): gastric infusion
  Interventions: Other: Infusion
- Duodenal (Experimental): Duodenal infusion
  Interventions: Other: Infusion

INTERVENTIONS:
Other: Infusion — infusion of nutrients

SUMMARY:
This pilot study will look at whether infusion of nutrients into the duodenum or into the stomach will result in:

1. decrease in hunger and food intake
2. greater weight loss due to loss of body fat with reductions in waist and hip circumferences
3. improvements in other weight-related health conditions such as diabetes, high blood pressure, and high blood triglycerides. Inclusion criteria: 25-60 years old with a BMI of ≥ 30≤55 kg/m2.

Subjects (16 individuals) will be in the study for 12 days and have a dobhoff tube placed at the start of the study. Subjects will visit MCRU daily for 12 days where meals will be provided, and where anthropometric measures, blood work during an oral mixed meal tolerance test (study start and study end), and surveys will be completed. The dobhoff tube will remain in place until the end of the study.

DETAILED DESCRIPTION:
The investigators propose a pilot study to evaluate whether mimicking rapid gastric emptying with duodenal infusion (DI) of nutrients (treatment) compared to gastric infusion (GI) of nutrients (control) over 12 days will result in 1) decrease in caloric intake 2) loss of body weight 3) improvements in comorbidities, particularly glucose metabolism, decrease in blood triglycerides and hypertension and increase in serum bile acids. Individuals eligible for the study will provide written informed consent. A comprehensive health and weight history will be obtained and physical exam obtained. Randomization will be 1:1 to DI vs. GI. There will be 8 individuals per treatment arm. A Dobhoff tube will be placed in each participant from nose either into duodenum (DI) or into stomach (GI). Participants will be allowed to eat three buffet style meals per day at 8.30 am, noon and 4 pm. The food intake will be noted for each meal by the investigators. Participants will note their feelings of hunger, fullness, bloating, nausea, and energy on a visual analogue scale every fifteen minutes for an hour starting at the initiation of the infusion. The placement of the tube (into stomach or duodenum) will be confirmed on day 1, day 6 and day 12 with radiographs. If necessary, fluoroscopy will be used only once during the study on day 1 to adjust the placement of the tube. During the study, the health of the participants will also be monitored and medications (if any) will be adjusted (if required) on a daily basis.

Intervention Group:

For first three days of the study (starting on Day#2), DI with 180 ml of warm saline will be given over 6 to 15 minutes through the Dobhoff tube starting a minute before initiation of each of the meal. For the remaining 7 days of the study, DI with nutrients in the form of 180 ml (266 Kcal) of warm Ensure Complete (Abbott Nutrition, OH) will be given over 6 to 15 minutes starting a minute before initiation of each meal. If they desire, participants will be allowed to eat a snack after the third meal.

Comparison group:

For first three days of the study (starting on Day#2), GI with 180 ml of warm saline will be given over 6 to 15 minutes through the Dobhoff tube starting a minute before initiation of each of the meal. For the remaining 7 days of the infusion part of the study, GI with nutrients in the form of 180 ml (266 Kcal) of warm Ensure Complete (Abbott Nutrition, OH) will be given over 6 to 15 minutes starting a minute before initiation of each meal. If they desire, participants will be allowed to eat a snack after the third meal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 25 and 60 years
* with body mass index (BMI) ≥30≤55 kg/m2

Exclusion Criteria:

* significant heart, kidney, liver, gastrointestinal tract (including gastrointestinal reflux disease), autoimmune disorders such as lupus erythematosus, neurological, psychiatric or endocrine disorders (Type 1 diabetes, adrenal, pituitary or uncontrolled thyroid disease), any previous surgeries on gastrointestinal tract, HIV/AIDS, anemia, clotting disorders, cancers other than minor skin cancers.
* individuals taking anti-obesity drugs, or appetite suppressants within the last 2 months.
* Individuals who have already undergone weight loss surgery are excluded.
* Women who intend to get pregnant, pregnant women and women who are nursing
* people who have a history of eating disorder such as bulimia or binge eating, or a history of or current substance abuse (alcohol, marijuana, cocaine, tobacco etc.).
* people who have stopped smoking within the previous 6 months and
* people with weight changes greater than 5 kg (about 11 pounds) within the previous 3 months.
* individuals who plan to move within 1 year.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12 days

SECONDARY OUTCOMES:
Change in body composition | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Amy Rothberg, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No